



## CT28-WI-GL01-RF01 2.0

# FINAL APPROVED PROTOCOL AND STATISTICAL ANALYSIS PLAN REDACTIONAPPROVAL FORM

31-Aug-2018

**PURPOSE:** This form is to be used by the approvers of the redacted final approved protocol (FAP) and/or statistical analysis plan (SAP) for public release. FAP and SAP approver signature denotes readiness for posting to ClinicalTrials.gov. and confirms intellectual property (IP) attorney review was completed.

### FAP AND/OR SAP REDACTION APPROVAL FORM

Protocol Number:

A0081105

Protocol Title:

A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center Trial of Pregabalin as Adjunctive Therapy in Pediatric and

Adult Subjects With Primary Generalized Tonic-Clonic Seizures -

Protocol -A0081105

Amendment Number (if

applicable):

N/A

Version Date:

26 July 2012

Phase:

3

SAP:

A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Trial of Pregabalin as Adjunctive Therapy in Pediatric and

Adult Subjects With Primary Generalized Tonic-Clonic Seizures

SAP Version Date:

18 March 2019

### FAP redaction approver

I have reviewed the redacted version of the FAP and confirm that it is appropriate for releasing publicly in accordance with global regulations and Pfizer policy.

☑ I confirm that IP has reviewed the redacted FAP.

**Print Name:** 

Signature: Lynne R Pauer

Date: 26 Jul 2019

08:10:057-0400

068f821f-a5ed-4065-b4e3-88d6f1d5beae

## SAP redaction approver

I have reviewed the redacted version of the SAP and confirm that it is appropriate for releasing publicly in accordance with global regulations and Pfizer policy.

#### PFIZER INTERNAL USE ONLY

The official version of this form is located in the electronic document management system and accessible via the eSOP portal.

Page 1 of 2



# CT28-WI-GL01-RF01 2.0

# FINAL APPROVED PROTOCOL AND STATISTICAL ANALYSIS PLAN REDACTIONAPPROVAL FORM

31-Aug-2018

| I confirm that IP has reviewed the redacted SAP. | | | 3 |
|--------------------------------------------------|-------|---------|---|
| Print Name: Rana Fayyad | | | |
| Signature: | Date: | 7/16/19 | |

## VERSION HISTORY

| Version | Effective Date | Change Type<br>(New, Revise,<br>Admin) | Summary of Revisions |
|---|---|---|---|
| 2.0 | 31-Aug-2018 | Admin | Administrative change - No new requirements added or process changes made. Clarified signatories and addresses minor inconsistencies with standard operating procedure (SOP) and added reminder that IP review is required according to the SOP. |
| 1.0 | 15-Feb-2018 | New | New form. |

### PFIZER INTERNAL USE ONLY

The official version of this form is located in the electronic document management system and accessible via the eSOP portal.